CLINICAL TRIAL: NCT04545008
Title: A Phase I Clinical Trial of the Combination of Famotidine (FAM) and Oral N-Acetyl Cysteine (NAC) Open Label for Outpatient Treatment of Subjects With Newly Diagnosed SARS-CoV-2 Infection
Brief Title: Trial of Famotidine & N-Acetyl Cysteine for Outpatients With COVID-19
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was stopped due to poor accrual.
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100394
Record Dates: First submitted 2020-09-01; First posted 2020-09-10 (Actual); Results first posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Covid19
Keywords: outpatient; famotidine; n-acetyl cysteine
MeSH Terms: conditions — COVID-19 | interventions — Famotidine; Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Low Dose N-Acetyl Cysteine Alone (Experimental): N-Acetyl Cysteine 600 mg three times daily
  Interventions: Drug: N-Acetyl cysteine
- Medium Dose N-Acetyl Cysteine (Experimental): N-Acetyl Cysteine 1,200 mg three times daily
  Interventions: Drug: N-Acetyl cysteine
- Low Dose N-Acetyl Cysteine and Low Dose Famotidine (Experimental): N-Acetyl Cysteine 600 mg three times daily Famotidine 20 mg three times daily
  Interventions: Drug: Famotidine; Drug: N-Acetyl cysteine
- High Dose N-Acetyl Cysteine Alone (Experimental): N-Acetyl Cysteine 1,800 mg three times daily
  Interventions: Drug: N-Acetyl cysteine
- Medium Dose N-Acetyl Cysteine and Low Dose Famotidine (Experimental): N-Acetyl Cysteine 1,200 mg three times daily Famotidine 20 mg three times daily
  Interventions: Drug: Famotidine; Drug: N-Acetyl cysteine
- Low Dose N-Acetyl Cysteine and Medium Dose Famotidine (Experimental): N-Acetyl Cysteine 600 mg three times daily Famotidine 40 mg three times daily
  Interventions: Drug: Famotidine; Drug: N-Acetyl cysteine
- High Dose N-Acetyl Cysteine and Low Dose Famotidine (Experimental): N-Acetyl Cysteine 1,800 mg three times daily Famotidine 20 mg three times daily
  Interventions: Drug: Famotidine; Drug: N-Acetyl cysteine
- Medium Dose N-Acetyl Cysteine and Medium Dose Famotidine (Experimental): N-Acetyl Cysteine 1,200 mg three times daily Famotidine 40 mg three times daily
  Interventions: Drug: Famotidine; Drug: N-Acetyl cysteine
- Low Dose N-Acetyl Cysteine and High Dose Famotidine (Experimental): N-Acetyl Cysteine 600 mg three times daily Famotidine 80 mg three times daily
  Interventions: Drug: Famotidine; Drug: N-Acetyl cysteine
- High Dose N-Acetyl Cysteine and Medium Dose Famotidine (Experimental): N-Acetyl Cysteine 1,800 mg three times daily Famotidine 40 mg three times daily
  Interventions: Drug: Famotidine; Drug: N-Acetyl cysteine
- Medium Dose N-Acetyl Cysteine and High Dose Famotidine (Experimental): N-Acetyl Cysteine 1,200 mg three times daily Famotidine 80 mg three times daily
  Interventions: Drug: Famotidine; Drug: N-Acetyl cysteine
- High Dose N-Acetyl Cysteine and High Dose Famotidine (Experimental): N-Acetyl Cysteine 1,800 mg three times daily Famotidine 80 mg three times daily
  Interventions: Drug: Famotidine; Drug: N-Acetyl cysteine

INTERVENTIONS:
Drug: Famotidine — Oral Famotidine
  Other Names: Pepcid AC
  Arms: High Dose N-Acetyl Cysteine and High Dose Famotidine; High Dose N-Acetyl Cysteine and Low Dose Famotidine; High Dose N-Acetyl Cysteine and Medium Dose Famotidine; Low Dose N-Acetyl Cysteine and High Dose Famotidine; Low Dose N-Acetyl Cysteine and Low Dose Famotidine; Low Dose N-Acetyl Cysteine and Medium Dose Famotidine; Medium Dose N-Acetyl Cysteine and High Dose Famotidine; Medium Dose N-Acetyl Cysteine and Low Dose Famotidine; Medium Dose N-Acetyl Cysteine and Medium Dose Famotidine
Drug: N-Acetyl cysteine — Oral N-Acetyl Cysteine
  Other Names: NAC

SUMMARY:
The purpose of this trial is to assess the safety and toxicity profile of the combination of famotidine and oral n-acetyl cysteine in adult outpatients with newly diagnosed SARS-CoV-2 infection.

DETAILED DESCRIPTION:
This is a phase I trial enrolling subjects with newly diagnosed SARS-CoV-2 infection who do not require hospitalization. Exclusion criteria have been written to exclude patients who would be expected to have increased risk from either medication alone. Subjects will be assigned a dose combination of famotidine and n-acetyl cysteine. In addition to assessing the safety and toxicities profiles of the combination of drugs we will be measuring certain endpoints to assess possible efficacy. These endpoint include the following: rates of hospitalization; time to complete remission of symptoms, e.g, fever, respiratory symptoms, etc.; severity of symptoms with validated survey instruments; cytokine values in serum and urine; and markers of inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* performance of a SARS-CoV-2 test within 1 day of enrollment, N.B., must be positive to proceed to treatment phase of the trial

Exclusion Criteria:

* All patients under 18
* Known allergy to N-Acetyl Cysteine
* Known allergy to famotidine or other H2-receptor antagonists
* Pregnant or Nursing Mothers
* Laboratory Evidence or History of Renal Impairment (eGFR < 30 mL/min/1.73 m2)
* Taking H2-receptor antagonists, hydroxychloroquine or chloroquine.
* Patient has been admitted to the hospital prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J O'Connell, M.D., Principal Investigator — Prisma Health
Locations (3):
- United States (3):
  - Prisma Health Baptist Easley Hospital, Easley, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Greer Memorial Hospital, Greer, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose N-Acetyl Cysteine Alone
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Dose N-Acetyl Cysteine Alone
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v5.0
Description: Data will be collected and entered into Case Report Form in local REDCap sever to include MedDRA Code, Grade and all other data required by NIH per Memorandum, "Guidance for Collection of Adverse Events Related to COVID-19 Infection" dated on 25 March 2020. All data will be reported per this memorandum and in accordance with all applicable Institutional Review Board and FDA requirements.
Time Frame: 0 to 30 days
Measure: Number; unit: participants
Arm/Group | Low Dose N-Acetyl Cysteine Alone
Number analyzed (Participants) | 2
participants | 0

2. Secondary Outcome: Rate of Hospitalization
Description: Number of participants hospitalized
Time Frame: 0 to 30 days
Measure: Number; unit: participants
Arm/Group | Low Dose N-Acetyl Cysteine Alone
Number analyzed (Participants) | 2
participants | 0

3. Secondary Outcome: Time to Symptom Resolution
Description: Days to resolution of symptoms of infection.
Time Frame: 0 to 30 days
Measure: Mean (Full Range); unit: days
Arm/Group | Low Dose N-Acetyl Cysteine Alone
Number analyzed (Participants) | 2
days | 6 [6 to 6]

ADVERSE EVENTS:
Time Frame: From consent to study completion, an average of 30 days.
Arm/Group | Low Dose N-Acetyl Cysteine Alone
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Decrease in COVID-19 infections in the area followed by other treatment options led to to poor enrollment (n=2) and early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT04545008/Prot_SAP_000.pdf